CLINICAL TRIAL: NCT01940640
Title: Multidisciplinary Study of the Effect of the Mother suplementación During the Lactation With High Doses of DHA on Diverse Aspects Related to the Development of the Premature Newborn in the First Year of Life.
Brief Title: Effect of Mother DHA Supplementation on Premature Newborn.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Julio J. Ochoa, Julio J. Ochoa, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AGL2011-24014
Record Dates: First submitted 2013-09-03; First posted 2013-09-12 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Oxidative Stress
Keywords: neonates, DHA
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA supplementation (Experimental): mothers consuming 900 mg DHA/day and their neonates.
  Interventions: Dietary Supplement: DHA
- Control (Active Comparator): follow on capsules without probiotics
  Interventions: Dietary Supplement: control

INTERVENTIONS:
Dietary Supplement: DHA — We will establish two groups of premature newborn children (<34 weeks) (n=40) and one group of newborn children to term (n=40). The mothers of one of the groups of premature newborn children will receive an oral supplementation by means of capsules with high dose of DHA (900 mg/day) during the lactation (minimum period of 3 months).
  Other Names: Docosahexaenoic acid
  Arms: DHA supplementation
Dietary Supplement: control — We will establish two groups of premature newborn children (<34 weeks) (n=40) and one group of newborn children to term (n=40). The mothers of one of the groups of premature newborn children will receive an oral supplementation by means of capsules with high dose of DHA during the lactation (minimum period of 3 months).
  Other Names: Follow on capsules without probiotics
  Arms: Control

SUMMARY:
To date, the investigations in the field of the supplementation with DHA in premature babies have been focused on the study of neuronal and visual development, giving place to contradictory and ambiguous results, because they did not consider in many cases important aspects of this supplementation, such as the mother´s diet, dose, duration, etc., and precise studies have not been performed in the field of the oxidative damage, inflammation and bone development in this population.

Hypothesis: If the composition of the mother´s milk is modified on the basis of her diet, a mother supplementation with high doses of DHA will increase proportionally the levels of this fatty acid in her milk, fact that will allows the premature newborn child receive a major dose of this fatty acid, and therefore this way, we will manage to improve the neuronal and visual development and to take part on the inflammatory process, oxidative damage and its evolution, together with the development or bone mass increase in the premature baby.

Aims: Overall we aim to evaluate in a multidisciplinary way the effect of a mother supplementation during the lactation with high doses of DHA on the development and wellness of the premature newborn children. We try to deepen into the effect on the neuronal and visual development and to study, for the first time, the effect on the oxidative damage, pro- and antiinflammatory citoquines activity and bone metabolism in this group of newborn babies.

DETAILED DESCRIPTION:
Experimental design: We will establish two groups of premature newborn children (<34 weeks) (n=40). The mothers of one of the groups of premature newborn children will receive an oral supplementation by means of capsules with high dose of DHA (900 mg/day) during the lactation (minimum period of 3 months). In addition, all the groups will be underwent to a nutritional surveillance (a follow-up of 48 hours and a questionnaire of frequency of consumption) and will be given nutritionally-balanced diets, insisting especially in the suitable consumption of fish (4 portions/week). Blood samples will be obtained in all the groups at the birth moment, at the week 40 of gestational age corrected in the groups of premature babies and at the end of the lactation in all the groups (minimum 3 months).We will obtain samples of mother´s milk (colostrum, transition and mature milk). In these samples we will study bone turnover biomarkers, pro - and anti-inflammatory citoquines and markers of aggression oxidative damage. In addition, we will perform psychomotor and visual development tests in the newborn children.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonate, gestational age 30-34, PAEG (>P10, <P95), no pathologies.

Exclusion Criteria:

* Lactose intolerance, systemic illness, multiple gestation, cromosomopathies, antibacterial therapy.

Ages: 1 Hour to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
blood and milk samples | at delivery
  Assessment of oxidative stress

SECONDARY OUTCOMES:
Blood | at delivery
  inflammation and bone development parameters

CONTACTS AND LOCATIONS:
Overall Officials: Julio J Ochoa, Ph.D., Principal Investigator — Universidad de Granada
Locations (1):
- Hospital San Cecilio, Granada, Granada, Spain